CLINICAL TRIAL: NCT02369263
Title: An Observational Study of Emergency Medicine Resident Performed Ultrasonography for DVT.
Brief Title: DVT Ultrasound in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Emergency Medicine Physicians, Nevada (Other)
Responsible Party: Sponsor
Other Study IDs: EMP2013-01
Record Dates: First submitted 2013-04-11; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Deep Vein Thrombosis; DVT
Keywords: Deep Vein Thrombosis; DVT; Leg Swelling; Leg Pain; Blood Clot
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Emergency Medicine (EM) Residents routinely conduct bedside ultrasound exams in the Emergency Department (ED) employing the two point compression method. This study endeavors to investigate the accuracy and utility of bedside ultrasound for Deep Vein Thrombosis (DVT) in the ED by EM Residents by comparing the results of that exam against the gold standard of a DVT ultrasound performed in the Radiology Department and interpreted by a Radiologist.

DETAILED DESCRIPTION:
For subjects with suspicion of DVT to the Emergency Department, an EM Resident will perform a bedside non-diagnostic two point compression DVT Ultrasound. Subjects will then receive a diagnostic DVT Ultrasound in the Radiology Department with official radiologist interpretation. The bedside ultrasound will not interfere with or delay the diagnostic ultrasound. Patient demographic and clinical data will be collected for validation purposes. Validation of the The EM Resident interpretation will be accomplished by comparison to the official Radiologist interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Suspect of having DVT

Exclusion Criteria:

* Known DVT
* DVT with in previous 6 months
* DVT Ultrasound within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Departmetn suspicious of DVT
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Outcome measures is the proportion of agreement between Resident performed two point DVT ultrasaound and the Radiologist interpertation of a formal DVT ultrasound. | 5 minutes
  Two point Emergency Medicine Resident preformed DVT Ultrasound (5 minute procedure) results will be compared as a proportion to Radiologist interpreted ultrasonographer performed DVT Ultrasound results.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Baydoun, MD, Principal Investigator — Emergency Medicine Physicians
Locations (1):
- University Medical Center of Southern Nevada, Las Vegas, Nevada, United States